CLINICAL TRIAL: NCT01044459
Title: A Long-Term, Randomized, Double-Blind Study of the Safety, Tolerability and Efficacy of Aclidinium Bromide At Two Dosage Levels When Administered to Patients With Moderate to Severe, Stable Chronic Obstructive Pulmonary Disease
Brief Title: Long-term Safety, Tolerability and Efficacy of Aclidinium Bromide in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) (LAS-MD-35)
Acronym: LAS-MD-35
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAS-MD-35
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium Bromide 200 µg (Experimental): aclidinium bromide, inhaled, 52 weeks of treatment
  Interventions: Drug: Aclidinium Bromide 200 µg
- Aclidinium Bromide 400 µg (Experimental): aclidinium bromide, inhaled, 52 weeks of treatment
  Interventions: Drug: Aclidinium Bromide 400 µg

INTERVENTIONS:
Drug: Aclidinium Bromide 200 µg — aclidinium bromide 200 μg, oral inhalation twice per day for 52 weeks of treatment
  Arms: Aclidinium Bromide 200 µg
Drug: Aclidinium Bromide 400 µg — aclidinium bromide 400 μg, oral inhalation twice per day for 52 weeks of treatment
  Arms: Aclidinium Bromide 400 µg

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of inhaled aclidinium bromide at two dose levels in patients with moderate to severe, stable chronic obstructive pulmonary disease. The study will be 56 weeks in duration; a 2-week rin-in period, a 52-week treatment period and a 2-week follow up phone call. All patients will be randomized to one of two doses of aclidinium bromide.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stable moderate to severe COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, 2010; postbronchodilator FEV1/FVC < 70%, and postbronchodilator FEV1 ≥ 30% and < 80% predicted
* Current or former cigarette smokers

Exclusion Criteria:

* Patients who have been hospitalized for an acute COPD exacerbation within 3 months before the first visit
* Respiratory tract infection or COPD exacerbation in the 6 weeks before Visit 1
* Patient with any clinically significant respiratory conditions other than COPD, cardiovascular conditions or mental illness
* History or presence of asthma verified from medical records
* Chronic use of oxygen therapy greater than or equal to 15 hours per day
* Patient with uncontrolled infection due to HIV and/or active hepatitis
* Patients with a history of hypersensitivity reaction to inhaled anticholinergics
* Patients with clinically significant cardiovascular conditions, including myocardial infarction during the previous 6 months, newly diagnosed arrhythmia within the previous 3 months, unstable angina, unstable arrhythmia that had required changes in pharmacological therapy or other intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (113):
- United States (110):
  - Forest Investigative Site 1162, Birmingham, Alabama
  - Forest Investigative Site 1127, Mobile, Alabama
  - Forest Investigative Site 1475, Scottsdale, Arizona
  - Forest Investigative Site 1338, Tempe, Arizona
  - Forest Investigative Site 1349, Tucson, Arizona
  - Forest Investigative Site 1483, Buena Park, California
  - Forest Investigative Site 1350, Foothill Ranch, California
  - Forest Investigative Site 1509, Fresno, California
  - Forest Investigative Site 2065, Fullerton, California
  - Forest Investigative Site 1502, Huntington Park, California
  - Forest Investigative Site 1088, Lakewood, California
  - Forest Investigative Site 1534, Long Beach, California
  - Forest Investigative Site 2209, Los Angeles, California
  - Forest Investigative Site 1122, Orange, California
  - Forest Investigative Site 1508, Palm Springs, California
  - Forest Investigative Site 2064, Riverside, California
  - Forest Investigative Site 1533, Sacramento, California
  - Forest Investigative Site 2009, San Diego, California
  - Forest Investigative Site 1439, San Diego, California
  - Forest Investigative Site 1503, San Diego, California
  - Forest Investigative Site 1347, San Jose, California
  - Forest Investigative Site 1344, Spring Valley, California
  - Forest Investigative Site 2039, Walnut Creek, California
  - Forest Investigative Site 2037, Fort Collins, Colorado
  - Forest Investigative Site 1327, Wheat Ridge, Colorado
  - Forest Investigative Site 1104, Hartford, Connecticut
  - Forest Investigative Site 1482, Stamford, Connecticut
  - Forest Investigative Site 1346, Newark, Delaware
  - Forest Investigative Site 1154, Brandon, Florida
  - Forest Investigative Site 1152, Clearwater, Florida
  - Forest Investigative Site 1514, Coral Gables, Florida
  - Forest Investigative Site 0670, DeLand, Florida
  - Forest Investigative Site 1516, Edgewater, Florida
  - Forest Investigative Site 0990, Fort Lauderdale, Florida
  - Forest Investigative Site 1513, Hialeah, Florida
  - Forest Investigative Site 1420, Miami, Florida
  - Forest Investigative Site 1432, Miami, Florida
  - Forest Investigative Site 1484, Miramar, Florida
  - Forest Investigative Site 1340, Ocala, Florida
  - Forest Investigative Site 1488, Pembroke Pines, Florida
  - Forest Investigative Site 0974, Pensacola, Florida
  - Forest Investigative Site 1397, Port Charlotte, Florida
  - Forest Investigative Site 1383, Port Orange, Florida
  - Forest Investigative Site 2082, Tamarac, Florida
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1395, Valrico, Florida
  - Forest Investigative Site 0980, Atlanta, Georgia
  - Forest Investigative Site 1491, Atlanta, Georgia
  - Forest Investigative Site 0987, Austell, Georgia
  - Forest Investigative Site 1532, Columbus, Georgia
  - Forest Investigative Site 2051, River Forest, Illinois
  - Forest Investigative Site 0989, Skokie, Illinois
  - Forest Investigative Site 1436, Avon, Indiana
  - Forest Investigative Site 2085, Crescent Springs, Kentucky
  - Forest Investigative Site 1520, Crestview Hills, Kentucky
  - Forest Investigative Site 0539, Lexington, Kentucky
  - Forest Investigative Site 1336, Louisville, Kentucky
  - Forest Investigative Site 1478, Louisville, Kentucky
  - Forest Investigative Site 2024, Lafayette, Louisiana
  - Forest Investigative Site 1333, Baltimore, Maryland
  - Forest Investigative Site 1421, Fall River, Massachusetts
  - Forest Investigative Site 1342, Stevensville, Michigan
  - Forest Investigative Site 1438, Ypsilanti, Michigan
  - Forest Investigative Site 2041, Minneapolis, Minnesota
  - Forest Investigative Site 1351, Plymouth, Minnesota
  - Forest Investigative Site 1100, Florissant, Missouri
  - Forest Investigative Site 2079, Saint Charles, Missouri
  - Forest Investigative Site 1343, St Louis, Missouri
  - Forest Investigative Site 1329, St Louis, Missouri
  - Forest Investigative Site 1369, St Louis, Missouri
  - Forest Investigative Site 1335, St Louis, Missouri
  - Forest Investigative Site 1367, Papillion, Nebraska
  - Forest Investigative Site 1150, Berlin, New Jersey
  - Forest Investigative Site 1339, Cherry Hill, New Jersey
  - Forest Investigative Site 1515, Elizabeth, New Jersey
  - Forest Investigative Site 1394, Ocean City, New Jersey
  - Forest Investigative Site 2062, Bronxville, New York
  - Forest Investigative Site 1147, Brooklyn, New York
  - Forest Investigative Site 1151, New Hyde Park, New York
  - Forest Investigative Site 1114, New York, New York
  - Forest Investigative Site 1163, New York, New York
  - Forest Investigative Site 1481, Newburgh, New York
  - Forest Investigative Site 0479, Rochester, New York
  - Forest Investigative Site 1368, The Bronx, New York
  - Forest Investigative Site 2081, Charlotte, North Carolina
  - Forest Investigative Site 1334, Charlotte, North Carolina
  - Forest Investigative Site 1366, HighPoint, North Carolina
  - Forest Investigative Site 1382, Statesville, North Carolina
  - Forest Investigative Site 1134, Canton, Ohio
  - Forest Investigative Site 2007, Cincinnati, Ohio
  - Forest Investigative Site 1434, Cleveland, Ohio
  - Forest Investigative Site 1433, Columbus, Ohio
  - Forest Investigative Site 0959, Columbus, Ohio
  - Forest Investigative Site 1505, Columbus, Ohio
  - Forest Investigative Site 1435, Dayton, Ohio
  - Forest Investigative Site 1348, Bend, Oregon
  - Forest Investigative Site 1504, Hershey, Pennsylvania
  - Forest Investigative Site 2072, Charleston, South Carolina
  - Forest Investigative Site 0900, Spartanburg, South Carolina
  - Forest Investigative Site 1365, Rapid City, South Dakota
  - Forest Investigative Site 0962, Nashville, Tennessee
  - Forest Investigative Site 1155, Dallas, Texas
  - Forest Investigative Site 1328, Dallas, Texas
  - Forest Investigative Site 1332, El Paso, Texas
  - Forest Investigative Site 1337, Houston, Texas
  - Forest Investigative Site 1396, San Antonio, Texas
  - Forest Investigative Site 1384, San Antonio, Texas
  - Forest Investigative Site 1330, South Burlington, Vermont
  - Forest Investigative Site 1120, Bellingham, Washington
  - Forest Investigative Site 1531, Tacoma, Washington
- Canada (3):
  - Forest Investigative Site 2201, Kelowna, British Columbia
  - Forest Investigative Site 1157, Toronto, Ontario
  - Forest Investigative Site 1168, Toronto, Ontario

REFERENCES:
- See also: las-md-35-synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4068&filename=las-md-35-synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from November of 2009 to April of 2010 at 109 study sites (106 sites in the United States and 3 additional sites in Canada). A total of 97 study sites randomized patients (94 in the United States and 3 in Canada).
Pre-assignment Details: A 2-week run-in period was used to assess the stability of patients' disease and to establish each patient's baseline characteristics. The run-in period was followed by a 52-week double-blind treatment period.
Groups:
- Aclidinium Bromide 200µg: Aclidinium bromide, 200 microgram dose, oral inhalation twice per day for 52 weeks of treatment.
- Aclidinium Bromide 400µg: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 52 weeks of treatment.
Period: Overall Study
Arm/Group | Aclidinium Bromide 200µg | Aclidinium Bromide 400µg
Started | 312 | 293
Completed | 179 | 162
Not Completed | 133 | 131
Not completed — Withdrawal by Subject | 21 | 28
Not completed — Terminated by Sponsor | 22 | 21
Not completed — Adverse Event | 22 | 20
Not completed — Lack of Efficacy | 23 | 12
Not completed — Protocol Violation | 11 | 16
Not completed — Other Reason | 7 | 14
Not completed — COPD exacerbation | 9 | 8
Not completed — Lost to Follow-up | 18 | 12

BASELINE CHARACTERISTICS:
Population: Of 605 patients randomized, 602 patients (99.5%) received at least 1 dose of double-blind treatment and were included in the Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide 200µg | Aclidinium Bromide 400µg | Total
Number analyzed (Participants) | 311 | 291 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (9.5) | 64.2 (9.9) | 63.6 (9.7)
Age, Customized [Number; unit: participants]
  ≥ 40 to < 60 years | 113 | 96 | 209
  ≥ 60 to < 70 years | 115 | 99 | 214
  ≥ 70 years | 83 | 96 | 179
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 124 | 251
  Male | 184 | 167 | 351
Region of Enrollment [Number; unit: participants]
  United States | 305 | 284 | 589
  Canada | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose (Trough) Forced Expiratory Volume in One Second (FEV1)
Description: Change From Baseline in Morning Predose (Trough) FEV1 in liters at Week 52.
Time Frame: From baseline to 52 weeks
Population: Of 605 patients randomized, 602 patients (99.5%) received at least 1 dose of double-blind treatment and were included in the Safety Population. Of these 602 patients, 600 (99.2%) had a baseline and at least 1 postbaseline FEV1 assessment and qualified for the ITT Population. A decision to terminate one site was made before unblinding of the study.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Aclidinium Bromide 200µg | Aclidinium Bromide 400µg
Number analyzed (Participants) | 310 | 290
L | 0.034 (0.015) | 0.072 (0.015)

2. Secondary Outcome: Change From Baseline in Peak FEV1
Description: Change From Baseline in Peak FEV1 in liters at Week 52.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Aclidinium Bromide 200µg | Aclidinium Bromide 400µg
Number analyzed (Participants) | 310 | 290
L | 0.185 (0.015) | 0.214 (0.015)

ADVERSE EVENTS:
Time Frame: Adverse event reporting occurred from November 2009 to May 2011 at 97 study sites (94 in the United States and 3 in Canada).
Description: Of 605 patients randomized, 602 patients (99.5%) received at least 1 dose of double-blind treatment and were included in the Safety Population; 311 patients for aclidinium bromide 200µg and 291 patients for aclidinium bromide 400µg
Arm/Group | Aclidinium Bromide 200µg | Aclidinium Bromide 400µg
Serious Adverse Events (participants affected / at risk) | 29/311 | 29/291
Other Adverse Events (participants affected / at risk) | 60/311 | 58/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 200µg (N=311) | Aclidinium Bromide 400µg (N=291)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Acute Myocardial Infarction (Cardiac disorders) | 2 | 2
Pneumonia (Infections and infestations) | 2 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cadiac Failure Congestive (Cardiac disorders) | 0 | 1
Carotid Artery Occlusion (Nervous system disorders) | 0 | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Clostridial Infection (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemophilus Infection (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Pharyngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia pneumococcal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Left atrial dilatation (Cardiac disorders) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermohypoaesthesia (Nervous system disorders) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 200µg (N=311) | Aclidinium Bromide 400µg (N=291)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 60 | 58

LIMITATIONS AND CAVEATS:
Site 1420 randomized 31 patients who were discontinued by 21 Jan 2011 due to significant deviations documented in a letter to the FDA on 07 Jan 2011. No changes to the analyses were prospectively specified in the amended statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.